CLINICAL TRIAL: NCT02669810
Title: EXpanded CELL ENdocardiac Transplantation (EXCELLENT)
Brief Title: EXCELLENT (EXpanded CELL ENdocardiac Transplantation)
Acronym: EXCELLENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CellProthera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT 2014-001476-63
Record Dates: First submitted 2016-01-25; First posted 2016-02-01 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PROTHERACYTES (Experimental): The interventional investigators will perform the ProtheraCytes® cardiac injections using a catheter introduced via the femoral route up to the left ventricle cavity for intraventricular injections (Helix/Biocardia).
  Intracoronary injection will be possible with OTW catheter or microcatheter (UK only) if patient presents a contraindication to intramyocardial injection
  Interventions: Drug: PROTHERACYTES; Drug: Standard Treatment for CHF post AMI
- Standard of Care (Active Comparator): Patients will be treated as standard treatment for CHF post - AMI.
  Interventions: Drug: Standard Treatment for CHF post AMI

INTERVENTIONS:
Drug: PROTHERACYTES — ProtheraCytes endocardiac injections performed with the HELIX and Morph catheters
  Arms: PROTHERACYTES
Drug: Standard Treatment for CHF post AMI

SUMMARY:
A multicentric controlled phase I / IIb study evaluating the safety and the efficacy of in vitro expanded peripheral blood CD34+ stem cells output by the StemXpand® Automated Process, and injected in patients with an acute myocardial infarction and a LVEF remaining below 50% versus standard of care.

DETAILED DESCRIPTION:
The main purpose of this phase I/IIb is to evaluate the safety, the tolerance and the first efficacy trends of intracardiac injection of ProtheraCytes (autologous PB-CD34+ Stem Cells after automated ex-vivo expansion with the StemXpand machine) in patients with an acute myocardial infarction and decreased ejection fraction. ProtheraCytes will be reinjected using a dedicated catheter , thus avoiding open chest surgery.

ELIGIBILITY:
Inclusion criteria

1. LV main AMI with or without ST segment elevation and with a detection of rise of troponin with at least one value 70 times above the upper reference limit.
2. MI within 1 week after first symptoms. D0 = day of last stent implantation or; D0 = day of hospital presentation when no stent implanted.
3. Combination of LVEF < 50% and LV akinetic or dyskinetic segment(s) - by echography as per local practice
4. Age must be ≥ 18 and ≤ 85 years
5. Men and Non-pregnant non-lactating women who take efficacious contraceptive measures such as oral contraceptive medications or efficacious and permanent intra-uterine device (drug eluted or not) (IUD) or subcutaneous permanent contraceptive implants or menopaused women (at least 2 years confirmed menopause) or surgically sterilized women.
6. Having previously signed a written informed consent prior to any study-specific procedure
7. LVEF remaining < 50% assessed by cMRI at D8 (± 3)
8. Identification of LV segment(s) both non-viable (transmural scar extend >50%) and akinetic (no cardiac wall thickening during systole) or dyskinetic (cardiac wall thickening in the wrong orientation during systole) by cMRI at D8 (± 3)

Non-inclusion criteria

1. History of CABG surgery
2. History of former significant mitral valve replacement surgery or heart transplantation.
3. History of severe valve disease: mitral, aortic stenosis / insufficiency.
4. History of non-ischemic dilated cardiomyopathy due to valvular dysfunction, mitral regurgitation, tachycardia, or myocarditis.
5. Aortic stenosis as determined as valve area less than 1 cm2 that prohibits catheter access to LV.
6. Presence of a prosthetic / mechanical aortic or mitral valve or heart constrictive device.
7. Sepsis.
8. Endocarditis.
9. Infectious pericarditis;
10. Pericardial tamponade.
11. Left Ventricular Thrombus detected at Echo or MRI
12. Severe peripheral vascular disease precluding femoral artery access as determined at the time of original catheterization.
13. Any condition leading to contraindicated or unexploitable cMRI.
14. History of metallic foreign body in their eye
15. Former or current aortic dissection
16. Previous G-CSF or other hematopoietic growth factor administration.
17. Hepatic failure, history of liver cirrhosis or hepatic severe impairment.
18. Constitutional or acquired coagulopathy
19. Treated chronic renal failure, haemodialysis or renal severe impairment (creatinine clearance < 30 ml/min).
20. Prior or concomitant malignancies except non-melanoma skin cancer or adequately treated in situ cervical cancer or previous cancer in complete response without any treatment in the last 5 years.
21. History of prior mediastinal radiation exposure.
22. Serious underlying medical condition at the investigator's discretion, which could impair the ability of the patient to participate in the trial (e.g. ongoing infection, active autoimmune disease, Amyotrophic Lateral Sclerosis, Systemic Lupus, Multiple Sclerosis).
23. Chronic immunomodulatory or cytotoxic drug treatment intake.
24. Active bleeding or major surgery within 1 month.
25. History or current Human immunodeficiency HIV1-2, HTLV1, HTLV2 (according to 2006/17/EC).
26. Current Active Hepatitis B (according to 2006/17/EC) based on the decision of the biologist or/and the PI.
27. History or current Hepatitis C (according to 2006/17/EC).
28. Syphilis (according to 2006/17/EC) based on the decision of the biologist or/and the P.
29. Active participation in any other clinical trials.
30. Current or recent treatment (within two months) with another investigational drug or procedure.
31. Any other co-existing conditions that will preclude participation in the study or compromise ability to give informed consent.
32. Impairment of cognitive function. If patient is 75-85 years old (included), score < 24 at Mini Mental State Examination (MMSE)
33. History of Splenomegaly;
34. History of Phenylketonuria;
35. History of iron-Dextran allergy;
36. History of murine protein allergy.
37. Diagnosis of Takotsubo

Discontinuation criteria

1. Inadequate bone marrow function: patient at risk to have Haemoglobin < 10 g/dL and Platelet count < 100 x 109 /L at the time of blood harvest
2. Blood transfusion within the previous 3 days before the first G-CSF injection
3. Cardiogenic shock: requirement of i.v. catecholamines or mechanical hemodynamic support (aortic balloon pump) initiated 24 hours before screening cMRI.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-09-25 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | From randomization up to 6 months
  The primary endpoint is the incidence of Major Adverse Cardiac Events (MACE), which have been adjudicated and confirmed to be a MACE by an independent and blinded Clinical Events Committee (CEC) from randomization

SECONDARY OUTCOMES:
Left Ventricle End Systolic Volume index (LVESVi) | From Baseline up to 6 months
  Improvement of LVESVi will be assessed by comparing cMRI at baseline, 3 and 6 months. The left ventricular volumes will be indexed to body surface area. cMRI will also assess other parameters such as:
  * Left ventricular end diastolic volume index (ml/m²)
  * Left ventricular ejection fraction (%)
  * Left ventricular mass (g)
Viability improvement of the infarcted segment(s) | From Baseline up to 6 months
  The viability assessment will be performed using cMRI and perfusion 99mTc SPECT (optional) respectively. A correlation assessment between LVESVi improvement and viability of the infarcted segment(s) will be statistically performed.
Other secondary outcomes measures | From Baseline up to 6 months
  Cardiac event free survival; Quality of life via SF36 scale

OTHER OUTCOMES:
Exploratory outcome measures | From randomization up to 6 months
  Incidence of adverse events in patient treated via the intracoronary route
Exploratory outcome measures | From randomization up to 6 months
  Improvement of MACE, of LVESVi, viability of infarcted segments and other cMRI parameters in patient treated with intracoronary route
Exploratory outcome measures | From Baseline up to 6 months
  cMRI parameters related to microvascular obstruction (MVO) and myocardial perfusion in all patients

CONTACTS AND LOCATIONS:
Locations (13):
- France (8):
  - CHU BESANCON Hopital Jean Minjoz 3 Boulevard A.Fleming, Besançon
  - CHU DIJON Hôpital François Mitterrand 14 rue Gaffarel, Dijon
  - CHU de Grenoble, Grenoble
  - Institut Jacques Cartier, Massy
  - CHU Montpellier Arnaud-De-Villeneuve, Montpellier
  - GHRMSA, Mulhouse
  - Hôpital Haut Levèque, Pessac
  - Hôpital de Rangueil, Toulouse
- United Kingdom (5):
  - Ninewells Hospital & Medical School, Dundee
  - BIRMINGHAM, Queen Elizabeth Hospital ,Mindelsohn Way,, Edgbaston
  - University of Edinburgh, Edinburgh
  - Leeds University & Leeds Teaching Hospitals NHS Trust, Leeds
  - Saint Bartholomew's Hospital W Smithfield,, London

REFERENCES:
- [Derived] Borlongan CV, Lee JY, D'Egidio F, de Kalbermatten M, Garitaonandia I, Guzman R. Nose-to-brain delivery of stem cells in stroke: the role of extracellular vesicles. Stem Cells Transl Med. 2024 Nov 12;13(11):1043-1052. doi: 10.1093/stcltm/szae072. PMID 39401332
- [Derived] Aries A, Vignon C, Zanetti C, Goubaud A, Cormier A, Diederichs A, Lahlil R, Henon P, Garitaonandia I. Development of a potency assay for CD34+ cell-based therapy. Sci Rep. 2023 Nov 11;13(1):19665. doi: 10.1038/s41598-023-47079-8. PMID 37952030